CLINICAL TRIAL: NCT06683573
Title: Optimizing Health Literacy and Disease Management Through 3D Kidney Model: Innovative Patient Education Approaches for Underserved Patients Impacted by Social Determinants of Health
Brief Title: Health Literacy 3D Kidney Model Patient Education Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hilary L Surratt, PhD (Other)
Collaborators: University of Kentucky (Other)
Responsible Party: Sponsor-Investigator, Hilary L Surratt, PhD, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 97260
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-01

CONDITIONS: High Blood Pressure; Kidney Disease, Chronic
MeSH Terms: conditions — Hypertension; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard clinical care/TAU (Active Comparator): standard clinician-led patient education
  Interventions: Behavioral: Standard medical treatment
- 3D Kidney model enhanced patient education (Experimental): patient education with 3D model
  Interventions: Behavioral: 3D Kidney model

INTERVENTIONS:
Behavioral: 3D Kidney model — Brief provider led counseling and education on Chronic Kidney Disease (CKD) and hypertension guided by use of 3D kidney model visual aid
  Arms: 3D Kidney model enhanced patient education
Behavioral: Standard medical treatment — Standard provider led counseling and education on CKD and hypertension
  Arms: Standard clinical care/TAU

SUMMARY:
High blood pressure has a different rate effect on many minoritized individuals. African Americans, as a result of high blood pressure, are six times more likely to go through kidney failure compared to white counterparts. Hispanic communities are also disproportionately affected by high blood pressure and, unfortunately, generally have lower knowledge about the effects on the kidneys as well. Unfortunately, many minoritized and underserved communities are affected by the weight of the social determinants of health, i.e., housing, education, food, health care, etc., that contribute to large disparities in health outcomes. These factors lead to poor care management, less ability to manage care effectively, and disengagement from care. Health education is vital to recognizing and communicating with minoritized patients with hypertension-induced chronic renal disease. As the patient's knowledge of the condition grows, this can significantly influence the trust between clinicians and patients. Effective and patient-centered education can inspire patients to be proactive in their prevention strategies with clinicians. This study's overall goal is to assess the utility of a novel patient education tool (3D-printed healthy kidney and diseased kidney models) in optimizing patient education for underserved populations who have hypertension with a potential lead to hypertension-induced chronic renal disease.

DETAILED DESCRIPTION:
The overall Aims of the study are to:

Aim 1: Examine the feasibility of creating a high-quality life-size 3D reconstruction of a healthy kidney model and diseased kidney model through collaboration with NIH 3D print exchange and the University of Kentucky College of Engineering.

Aim 2: Assess the acceptability and preliminary efficacy of 3D print model-supported patient education in improving the patients' medical understanding, motivation for self-care, intention to adhere to the clinician's instructions, and better trust between clinician and patient.

Aim 3: Continuously implement of 3D-printed models for patients in new or current care education so that it can be sustainable after the research project is concluded.

To achieve Aim 2, up to 100 patients with hypertension-induced chronic renal disease will be enrolled and randomized to receive either standard clinician-led patient education (TAU) or patient education employing the 3D kidney model. A brief pre-post structured survey will be implemented to measure changes in patients' understanding of their condition, as well as acceptability of the 3D model for those assigned to the experimental education condition.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 and older
* Seeking medical care in study location
* Current diagnosis of hypertension and renal disease

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2025-02-25 (Actual); Primary Completion 2025-03-27 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
Change in participant confidence for kidney disease management | Baseline and post intervention, approximately 1 hour
  Participant confidence will be measured by a survey with a Likert type scale where higher scores equate to increased confidence.

CONTACTS AND LOCATIONS:
Overall Officials: Hilary L Surratt, PhD, Study Chair — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No